CLINICAL TRIAL: NCT07257302
Title: Exploratory Study on the Effects of Lung Insufflation Capacity Training Using the LIC Trainer in Patients With Amyotrophic Lateral Sclerosis: A Single-Center Prospective Interventional Study
Brief Title: Lung Insufflation Capacity Training and Respiratory Function in Amyotrophic Lateral Sclerosis
Acronym: LIC-ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Principal Investigator, Taiyo Kawaguchi, Physician, Department of Rehabilitation Medicine, National Center of Neurology and Psychiatry, Japan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCNP-LIC-ALS-2025; 25K14423 (Other Grant/Funding Number: Japan Society for the Promotion of Science (JSPS))
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: LIC Trainer; lung volume recruitment; respiratory rehabilitation; FVC; ALS; ALSFRS-R; cough peak flow
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Single-arm prospective study comparing pre- and post-intervention changes in respiratory function among patients with ALS receiving LIC training.
Masking Description: All participants and investigators are aware of the intervention. No blinding is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LIC Training (Experimental): Participants with amyotrophic lateral sclerosis (ALS) will perform lung insufflation capacity (LIC) training using the LIC Trainer device to maintain lung and chest wall compliance. Each session consists of about 10 assisted insufflations performed twice daily at home. Physical therapists provide initial instruction and re-evaluation every 3 months during the 36-month follow-up period. The intervention aims to preserve pulmonary function, reduce respiratory complications, and prolong survival.
  Interventions: Device: LIC Trainer (Lung Insufflation Capacity Trainer)

INTERVENTIONS:
Device: LIC Trainer (Lung Insufflation Capacity Trainer) — The LIC Trainer is a medical device designed to enable lung insufflation through a one-way valve system, allowing passive air stacking without voluntary glottic closure. The device includes a safety valve that automatically releases pressure above 60 cmH₂O and a manual relief valve to ensure patient safety. It is used with a bag-valve-mask to deliver multiple assisted insufflations, approximately 10 per session, twice daily. Participants with amyotrophic lateral sclerosis (ALS) perform LIC training at home after initial instruction by physical therapists and are re-evaluated every 3 months for up to 36 months.
  Other Names: Lung Insufflation Capacity Trainer; LIC training; air stacking training

SUMMARY:
The goal of this clinical trial is to learn whether lung insufflation capacity (LIC) training can help maintain respiratory function and prolong survival in people with amyotrophic lateral sclerosis (ALS).

The main questions it aims to answer are:

* Does early and continuous LIC training slow the decline in forced vital capacity (FVC)?
* Does LIC training delay the need for tracheostomy or noninvasive ventilation (NIV)? This single-center study at the National Center of Neurology and Psychiatry (NCNP) in Japan will enroll 15 adults with ALS, diagnosed according to the El Escorial or Awaji criteria.

Participants will:

* Use the LIC Trainer device to perform lung insufflation training twice daily at home
* Visit the clinic every 3 months for respiratory and functional assessments
* Have lung tests, including FVC, LIC, maximum insufflation capacity (MIC), cough peak flow (CPF), and complete the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) There is no control group within this trial; researchers will compare results with matched historical controls from the Pooled Resource Open-Access ALS Clinical Trials (PRO-ACT) database.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease characterized by upper and lower motor neuron degeneration, leading to muscle weakness, functional decline, and ultimately respiratory failure. Respiratory muscle weakness causes restrictive ventilatory impairment and a progressive decrease in forced vital capacity (FVC), which is strongly associated with survival. Because no curative therapy exists, respiratory rehabilitation aimed at maintaining pulmonary function and chest wall compliance plays an important role in extending quality of life and survival.

Lung volume recruitment therapy (LVRT) is a respiratory rehabilitation method that uses assisted lung inflation to expand the lungs and maintain compliance. It is commonly performed with a manual resuscitation bag (bag-valve-mask, BVM) by stacking multiple breaths to reach maximum insufflation capacity (MIC). However, this conventional method requires voluntary glottic closure to maintain air stacking. In people with ALS who have bulbar symptoms or tracheostomy, this ability is often lost, making conventional LVRT difficult or impossible.

To overcome this limitation, a device-based approach known as lung insufflation capacity (LIC) training was developed. The LIC Trainer is a licensed medical device in Japan that allows air stacking through a one-way valve mechanism, enabling passive insufflation without voluntary glottic control. The device incorporates a safety valve that automatically opens at pressures above 60 cmH₂O to prevent barotrauma and a manual relief valve allowing patient-controlled exhalation. Although the LIC Trainer has been used clinically in Japan since 2016, evidence regarding its long-term effects in ALS remains limited.

This prospective single-center interventional study aims to evaluate the effects of LIC training on respiratory function and survival in adults with ALS at the National Center of Neurology and Psychiatry (NCNP), Tokyo, Japan. Participants are diagnosed with ALS according to the El Escorial or Awaji criteria, are 20 years of age or older, and are not using noninvasive ventilation (NIV) and do not have a tracheostomy at the start of LIC training. Key exclusion criteria include other chronic pulmonary diseases, severe cardiac dysfunction, and conditions that preclude study assessments.

After providing written informed consent, participants receive education on LIC training from a physical therapist and are provided with an LIC Trainer and bag-valve-mask for home use. They are instructed to perform a set of insufflation cycles, typically around 10 per session, twice daily. Training logs are maintained by participants and reviewed at each visit to monitor adherence and safety. Outpatient follow-up visits occur every 3 months for up to 36 months.

At each visit, respiratory function (percent predicted FVC, LIC, MIC, cough peak flow [CPF], and assisted CPF) and functional status (Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised [ALSFRS-R]) are assessed. Clinical events such as respiratory infections, hospitalizations, tracheostomy, and death are also recorded. The primary outcome is overall survival, defined as the time from initiation of LIC training to tracheostomy or death. Secondary outcomes include longitudinal changes in respiratory function and ALSFRS-R scores, as well as the frequency of respiratory infections.

Data from this intervention group will be compared with a matched historical control cohort derived from the Pooled Resource Open-Access ALS Clinical Trials (PRO-ACT) database. Propensity score matching will be used to balance baseline characteristics such as age, sex, site of onset, percent predicted FVC, body mass index (BMI), ALSFRS-R, and use of riluzole and edaravone. Survival will be analyzed using Kaplan-Meier estimates and Cox proportional hazards models, and repeated measures of respiratory and functional outcomes will be analyzed using linear mixed-effects models. This study is expected to clarify whether early and sustained LIC training can help maintain lung and chest wall compliance, slow the decline in respiratory function, and potentially extend survival in ALS.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older
* Diagnosis of amyotrophic lateral sclerosis (ALS) according to the El Escorial or Awaji criteria
* Not using noninvasive ventilation (NIV) and without tracheostomy at the start of LIC training
* Able to perform study assessments and provide written informed consent (or assisted signature with communication aid)

Exclusion Criteria:

* Chronic pulmonary disease other than ALS (e.g., COPD, interstitial lung disease)
* Severe cognitive or communication impairment preventing study participation
* Uncontrolled cardiovascular disease, including unstable angina, recent myocardial infarction, decompensated heart failure, serious arrhythmia, severe aortic stenosis, or active myocarditis/endocarditis
* Uncontrolled hypertension
* Acute systemic illness or fever
* Recent pulmonary embolism, acute cor pulmonale, or severe pulmonary hypertension
* Severe hepatic or renal dysfunction
* Any condition judged inappropriate by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (time to tracheostomy or death) | From the start of LIC training (Day 0) until tracheostomy or death, up to 36 months
  Overall survival is defined as the time from the initiation of lung insufflation capacity (LIC) training to tracheostomy or death, whichever occurs first. Participants who remain alive without tracheostomy at the end of follow-up will be censored at their last known assessment. Survival analysis will use Kaplan-Meier estimates and Cox proportional hazards models. The outcome will also be compared with matched historical controls from the PRO-ACT ALS database using propensity score matching.

SECONDARY OUTCOMES:
Change in forced vital capacity (%FVC) | Baseline and every 3 months for up to 36 months
  Forced vital capacity (FVC, expressed as percent predicted) will be measured every 3 months to assess longitudinal respiratory function. The rate of decline in %FVC before and after initiation of LIC training will be compared using linear mixed-effects models.
Change in lung insufflation capacity (LIC) and maximum insufflation capacity (MIC) | Baseline and every 3 months for up to 36 months
  LIC and MIC will be assessed at each visit using the LIC Trainer and bag-valve-mask method, respectively. The difference between LIC or MIC and FVC (LIC-FVC, MIC-FVC) will also be evaluated to determine lung and chest wall compliance over time.
Change in cough peak flow (CPF) and assisted CPF | Baseline and every 3 months for up to 36 months
  Peak cough flow (CPF) and assisted CPF will be measured using a spirometer to evaluate expiratory muscle strength and effectiveness of airway clearance. Longitudinal changes will be analyzed using mixed-effects models.
Change in ALS Functional Rating Scale-Revised (ALSFRS-R) score | Baseline and every 3 months for up to 36 months
  Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) total and subscale scores (bulbar, limb, and respiratory domains) will be assessed to evaluate overall disease progression. The ALSFRS-R is a 12-item scale with total scores ranging from 0 to 48, where higher scores indicate better functional status and lower scores indicate more severe disability. The monthly slope of ALSFRS-R decline will be calculated and compared with matched historical controls.
Incidence of respiratory infections | Up to 36 months
  Respiratory infection events (e.g., pneumonia) will be recorded, including onset date, hospitalization, and antibiotic use. Annualized event rates will be compared before and after LIC training using Poisson or negative binomial regression, and time to first infection will be analyzed with Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Taiyo Kawaguchi, MD, Principal Investigator — National Center of Neurology and Psychiatry
Locations (1):
- National Center of Neurology and Psychiatry (NCNP), Kodaira, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared outside the study team due to ethical and regulatory constraints. Summary data and study findings may be made available in publications or upon reasonable request.

REFERENCES:
- See also: Public registration record in the UMIN Clinical Trials Registry (Japan) — https://center6.umin.ac.jp/cgi-open-bin/ctr_e/ctr_view.cgi?recptno=R000067849